CLINICAL TRIAL: NCT01397084
Title: An 8-week, Open Label, Multicentre Study to Assess the Efficacy of Esomeprazole 20 mg Once Daily in Subjects With Continuing Symptoms of Heartburn Following Treatment With a Previous Rabeprazole
Brief Title: To Assess the Efficacy of Esomeprazole 20mg Once Daily in Subjects Who Still Had Heartburn After Receiving Rabeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D961HL00002
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Reflux Esophagitis
Keywords: esomeprazole 20mg; heartburn; rabeprazole 10mg; reflux esophagitis; Phase IV
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic; Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- esomeprazole 20 mg (Other): esomeprazole 20 mg
  Interventions: Drug: esomeprazole 20 mg

INTERVENTIONS:
Drug: esomeprazole 20 mg — esomeprazole 20 mg once daily for 8 weeks

SUMMARY:
Administration of esomeprazole 20 mg to subjects who still had heartburn after receiving rabeprazole 10 mg once daily for at least 4 weeks will result in statistically significant improvement of heartburn after 8-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male of female aged 20 years or more
* History of reflux esophagitis
* Ongoing (until date of Visit 1) treatment with rabeprazole 10 mg, given once daily, for at least 4 weeks.The subject must take rabeprazole at least 4 days a week in the past 7 days prior to Visit 1.
* Persisting symptoms of heartburn experienced at least 2 days during the past 7 days prior to Visit 1.

Exclusion Criteria:

* Use of other PPIs and/or H2RA during rabeprazole treatment
* History or having other gastrointestinal diseases
* History of upper gastrointestinal surgery
* Initiation of medications that can affect digestive functions within 4 weeks before study treatment
* Inability to complete questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, Study Director — AZ K.K.; Makiko Abe, Study Chair — AZ K.K

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on 25 August 2011. Last participant completed on 31 January 2012. Out of 108 enrolled participants, 107 participants (target was 100) received esomeprazole 20 mg. All of the participants were included in safety analysis set and 104 out of the 107 participants were included in the full analysis set for efficacy analyses.
Pre-assignment Details: Participants with a history of reflux oesophagitis and with continuing heartburn after previous treatment with rabeprazole 10 mg were included in this study.
Groups:
- Esomeprazole 20 mg: esomeprazole 20 mg : esomeprazole 20 mg once daily for 8 weeks
Period: Overall Study
Arm/Group | Esomeprazole 20 mg
Started | 108
Completed | 100
Not Completed | 8
Not completed — Severe Non-Compliance to Protocol | 1
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Used other proton pump inhibitor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esomeprazole 20 mg
Number analyzed (Participants) | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of Heartburn During the 7-day Period Prior to the 8 Week Visit (Visit 3) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1).
Description: The number of days with heartburn during the 7-day period prior to the 8 week visit (Visit 3) was compared to the number of days with heartburn during the 7-day period prior to baseline (Visit 1). The difference in the number of days with heartburn from baseline to 8 weeks was analysed.
Time Frame: Baseline and 8 weeks
Population: Efficacy Population (104 participants)
Measure: Mean (Standard Deviation); unit: Days with heartburn
Arm/Group | Esomeprazole 20 mg
Number analyzed (Participants) | 104
Days with heartburn | -3.0 (2.4)
Statistical Analysis 1: Comparison: Esomeprazole 20 mg; Wilcoxon signed-rank test was used to check whether the change in the frequency of heartburn during the 7-day period prior to the 8 week visit (Visit 3) compared to the frequency of heartburn during the 7-day period prior to baseline (Visit 1) was statistically significant or not; Test type: Superiority or Other; p < 0.001, Wilocoxon signed-rank test

2. Secondary Outcome: Change in the Frequency of Heartburn During the 7-day Period Prior to the 4 Week Visit (Visit 2) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1).
Description: The number of days with heartburn during the 7-day period prior to the 4 week visit (Visit 2) was compared to the number of days with heartburn during the 7-day period prior to baseline (Visit 1). The difference in the number of days with heartburn from baseline to 4 weeks was analysed.
Time Frame: Baseline and 4 weeks
Population: 101 Participants out of efficacy population (104 participants) who had data related to heartburn at Week 4 were used.
Measure: Mean (Standard Deviation); unit: Days with heartburn
Arm/Group | Esomeprazole 20 mg
Number analyzed (Participants) | 101
Days with heartburn | -2.4 (2.8)

3. Secondary Outcome: Change in the Maximum Severity of Heartburn During the 7-day Period Prior to the 4 Week Visit (Visit 2) Compared to the Maximum Severity of Heartburn During the 7-day Period Prior to Baseline (Visit 1).
Description: Maximum severity of heartburn during 7 days at baseline and at 4 weeks was obtained (None, Mild, Moderate, Severe). If the value at 4 weeks was better than at baseline in a participant, the participant was s categorized into "Improved". If the value was same, then categorised into "Unchanged". If the value was worsened, categorised into "Worsened".
Time Frame: Baseline and 4 weeks.
Population: 101 Participants out of efficacy population (104 participants) who had data related to heartburn at Week 4 were used.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20 mg
Number analyzed (Participants) | 101
Participants
  Improved | 76
  Unchanged | 24
  Worsened | 1

4. Secondary Outcome: Change in the Maximum Severity of Heartburn During the 7-day Period Prior to the 8 Week Visit (Visit 3) Compared to the Maximum Severity of Heartburn During the 7-day Period Prior to Baseline (Visit 1).
Description: Maximum severity of heartburn during 7 days at baseline and at 8 weeks was obtained (None, Mild, Moderate, Severe). If the value at 8 weeks was better than at baseline in a participant, the participant was s categorized into "Improved". If the value was same, then categorised into "Unchanged". If the value was worsened, categorised into "Worsened".
Time Frame: Baseline and 8 weeks
Population: Efficacy Population (104 participants)
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20 mg
Number analyzed (Participants) | 104
Participants
  Improved | 84
  Unchanged | 18
  Worsened | 2

ADVERSE EVENTS:
Arm/Group | Esomeprazole 20 mg
Serious Adverse Events (participants affected / at risk) | 2/107
Other Adverse Events (participants affected / at risk) | 2/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20 mg (N=107)
Typhoid Fever (Infections and infestations) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20 mg (N=107)
Diarrhoea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.